CLINICAL TRIAL: NCT05881083
Title: Building Capacity and Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2023: a Randomised Controlled Trial of 1-week Nicotine Replacement Therapy Sampling
Brief Title: Nicotine Replacement Therapy Sampling for Smokers in the Community
Acronym: QTW2023
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Principal Investigator, Tzu Tsun Luk, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QTW2023
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Tobacco Smoking
Keywords: smoking; tobacco; nicotine replacement therapy; lay counsellor
MeSH Terms: conditions — Tobacco Smoking; Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 1-week nicotine replacement therapy sample + Brief cessation advice
  Interventions: Behavioral: 1-week nicotine replacement therapy sampling; Behavioral: Brief cessation advice
- Control group (Active Comparator): Brief cessation advice
  Interventions: Behavioral: Brief cessation advice

INTERVENTIONS:
Behavioral: 1-week nicotine replacement therapy sampling — Participants will be given an 1-week sample of nicotine replacement therapy (patch or gum) with brief instructions on how to use the product
  Arms: Intervention group
Behavioral: Brief cessation advice — Participants will receive brief cessation advice following the AWARD (ask, warn, advise, refer, do-it-again) model:
  A: Ask about the tobacco use status; W: Warn about the hazards of tobacco use; A: Advise the smokers to quit; R: Refer the smokers to cessation services; D: Do-it-again

SUMMARY:
The aim of this clinical trial is to test the effectiveness of 1-week nicotine replacement therapy sampling delivered by lay counsellors in promoting smoking cessation in smokers in the community.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged 18 years or above
2. Smoke cigarette or heated tobacco product or e-cigarette daily in the past 3 months
3. Exhaled carbon monoxide level ≥4 part per million or a positive salivary cotinine test
4. Able to communicate in and read Chinese
5. Have a local contact number

Exclusion Criteria:

1. Participating in another smoking cessation programme or using any smoking cessation drug or nicotine replacement therapy
2. Pregnant or breastfeeding
3. Recent (≤ 2 weeks) angina, cardiac arrhythmia or heart attacks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1014 (Estimated)
Dates: Start 2023-06-17 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated tobacco abstinence | 6 months
  Verified by a negative salivary cotinine test

SECONDARY OUTCOMES:
Biochemically validated tobacco abstinence | 3 months
  Verified by a negative salivary cotinine test
Self-reported 7-day point-prevalence tobacco abstinence | 3 months
Self-reported 7-day point-prevalence tobacco abstinence | 6 months
Self-reported 24-hour quit attempt | 3 months
Self-reported 24-hour quit attempt | 6 months
Self-reported use of nicotine replacement therapy product | 3 months
Self-reported use of nicotine replacement therapy product | 6 months
Self-reported use of smoking cessation service | 3 months
Self-reported use of smoking cessation service | 6 months

OTHER OUTCOMES:
Self-reported reduction of tobacco consumption | 3 months
  Smoking reduction by at least half of the baseline daily number of cigarettes
Self-reported reduction of tobacco consumption | 6 months
  Smoking reduction by at least half of the baseline daily number of cigarettes
Change in motivation to quit from baseline through 3-month follow-up | 3 months
Change in motivation to quit from baseline through 6-month follow-up | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tzu Tsun Luk, PhD, RN, Principal Investigator — The University of Hong Kong
Locations (1):
- Community sites, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No